CLINICAL TRIAL: NCT05033600
Title: Low-Voltage, Direct Current Pulsed ElectroMagnetic Field (PEMF) Therapy in Treating Patients With Post-Traumatic Stress Disorder (PTSD and cPTSD) and Trauma
Brief Title: Pulsed ElectroMagnetic Field (PEMF) Therapy in Treating Post-Traumatic Stress Disorder (PTSD) & Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasey Phifer (Other)
Collaborators: The National Centre for ElectroMagnetic Therapies CIC (Other)
Responsible Party: Sponsor-Investigator, Kasey Phifer, Director & Lead Practitioner, The National Centre for ElectroMagnetic Therapies CIC
Organization: The National Centre for ElectroMagnetic Therapies CIC (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTSD-Trauma-PEMF-PS2021
Record Dates: First submitted 2021-07-20; First posted 2021-09-05 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Unspecified Trauma- and Stressor-Related Disorder
Keywords: PTSD; cPTSD; Anxiety; Insomnia; Self-Sabotage; Hyper-Sensitivity; Flashbacks; Irritability
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This pilot study has one arm only: PEMF therapy treatment. This pilot study does not make use of a placebo, no double-blind, and no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional - PEMF Therapy Recipients (Experimental): 90-minute sessions rendered twice weekly over three consecutive weeks. PEMFs are administered through electrodes attached to wrists, ankles and forehead of participant.
  Interventions: Device: S.C.I.O.

INTERVENTIONS:
Device: S.C.I.O. — The devices read, emit and entrain Electromagnetic waves of the body.
  Other Names: Scientific Consciousness Interface Operations Biofeedback Device; Nucleus Device; Eductor Device; Eductor1 Device

SUMMARY:
Use of low-voltage, direct current pulsed electromagnetic fields (PEMF) in treating Post Traumatic Stress Disorder (PTSD), complex PTSD (cPTSD) and trauma-related injuries manifesting in physical and/or mental symptoms.

DETAILED DESCRIPTION:
The PEMF devices used are the Scientific Consciousness Interface Operations (SCIO) device; it is CE-marked, ISO certified and FDA classified as a Type II medical device. The device measures frequencies emitted by the patient as a Biofeedback tool, and then emits frequencies in square (50% duty cycle), sinus or sawtooth wave form.

Wave forms, frequencies (herz and kiloherz respectively), ampers and voltage are adjusted automatically using the in-built Artificial Intelligence of the software employed to control the SCIO machine. The maximum is 5 Direct Current volts.

Electrodes to both read and emit signals are placed on the forehead, wrists and ankles. Irregular frequencies are corrected by use of entrainment. Efficacy of entrainment is displayed in the software as a percentage between 0-100. A rectification level or entrainment result of 85-100% is considered successful treatment, that is, entrainment was as effective as possible for that one session.

PEMF therapy has already been shown to be effective in trauma, PTSD, anxiety and depression treatment. The University of Denmark have recently conducted a similar clinical trial, which investigated Transcranial Direct Current Electro-Magnetic Therapy for patients who were treatment-resistant to depression medication. This study was also a one-arm test. This test was conducted over the space of 8 weeks and involved 52 participants of mixed gender. All the results indicated a reduction in depression-related symptoms in different ways, using the Hamilton Depression Scale as a reference point. The baseline of the Hamilton Depression Scale dropped from 20.6 to 12.6, whilst 49 participants experienced a reduction of over 50% on the Hamilton Depression Scale. Their study concluded that Transcranial Electro-Magnetic Therapy was a beneficial treatment for treatment-resistant depression, and further studies should be conducted to highlight the potential benefits of similar treatments.

This pilot study does not make use of a placebo, no double-blind, and no control group. The aim of this pilot study is two-fold: Firstly to determine whether a lower total amount of sessions would be effective (namely twice weekly rather than five days a week over the course of three weeks); secondly, whether the setup and process of this pilot study can function at scale (multiple locations and relatively little training time required by therapists due to the artificial intelligence built into the software guiding the machine).

ELIGIBILITY:
Inclusion Criteria:

* Human adults above or equal to 19 years of age
* All sexes and genders
* It is okay if they are currently seeking or undergoing complementary therapies and treatments for their PTSD such as cognitive behavioural therapy or anti-depressant pharmaceutical medications
* Diagnosed with PTSD and/or trauma
* Experiencing symptoms of PTSD and/or trauma, listed below:
* Re-imagining or 3D flash backs
* Sudden bouts of anger or irritability
* Self-sabotage
* Reliance upon coping mechanisms such as drugs or alcohol
* Insomnia
* Hyper-sensitivity
* Anxiety
* Able to travel to one of 3 treatment locations in London, Bristol or Bournemouth at the participant's own expense
* Able to attend all 6 treatments consisting of twice-weekly therapy sessions each 90 minutes in duration for three consecutive weeks

Exclusion Criteria:

* Any person on medication for severe psychotic episodes and/or suicidal thoughts / attempts
* Anyone under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Anxiety | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.
Hyper-Sensitivity | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.
Insomnia | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.
Self-Sabotage | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.
Reliance upon coping mechanisms such as drugs or alcohol | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.
Re-imagining or 3D flash backs | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.
Sudden outbursts of anger, mood swings, irritability | 3 weeks
  We will have a questionnaire for all patients. This will include ratings of their mood and feelings related to each of these symptoms. This questionnaire will be used in comparison to a similar questionnaire completed prior to the start date of the clinical trial. Rating systems such as 1 to 10 will be used, as well as an opportunity to write freely about their experiences during the trial. Statements will be used in which patients reply their own thoughts to them.

CONTACTS AND LOCATIONS:
Overall Officials: Kasey Phifer, B.A., Study Director — The National Centre for ElectroMagnetic Therapies CIC
Locations (1):
- The National Centre for ElectroMagnetic Therapies CIC - Private Clinic at Hillside Studios, Berwick Lane, Easter Compton, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
anonymised data will be shared in raw format (spreadsheet .csv), analysed data will be disseminated first-hand and through peer-reviewed channels
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data should be made available in October 2021 on the company website
Access Criteria: No access criteria, publicly available
URL: https://ncet.co.uk

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT05033600/Prot_SAP_000.pdf